CLINICAL TRIAL: NCT06129136
Title: The Effect of Nature-based Exposure on the Immune System and Skin Health of Atopic Dermatitis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uute Scientific Oy (Industry)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Uuteatopia2
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
Keywords: Biodiversity intervention; Allergy; Atopy; Environmental microbes
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are randomized to groups by external statistician. Test lotions are looking the same so participants and investigators don't know in which group they are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nature-based exposure by biodiversity component in lotion. (Active Comparator): This group uses regularly the lotion with added natural biodiversity component. The component is mimicking natural exposure to Finnish forest soil and it contains high microbial diversity. The microbes are inactivated.
  Interventions: Other: Nature-based exposure by biodiversity component in lotion.
- Placebo group using colored lotion. (Placebo Comparator): This group uses regularly the same vehicle lotion than Nature exposure group, with the difference that the biodiversity component has been replaced with safe coloring ingredients to give the same brownish color than in the other group's lotion. Coloring ingredients are iron oxides that are common in foods and cosmetics: C.I.7791, C.I.77492, C.I. 774499.
  Interventions: Other: Placebo group using colored lotion.

INTERVENTIONS:
Other: Nature-based exposure by biodiversity component in lotion. — Lotion is used at minimum three times per week and at least to arms. No restrictions to normal life and self-care. Atopy medicines and lotions are allowed when needed, only the usage amount is followed.
  Arms: Nature-based exposure by biodiversity component in lotion.
Other: Placebo group using colored lotion. — Lotion is used at minimum three times per week and at least to arms. No restrictions to normal life and self-care. Atopy medicines and lotions are allowed when needed, only the usage amount is followed.
  Arms: Placebo group using colored lotion.

SUMMARY:
The purpose of the study is to explore the effect of nature-based exposure on immunological biomarkers and the condition and symptoms of atopic skin. Our hypothesis is that regular exposure to nature-based, high biodiversity material on skin, strengthens the skin's protective barrier and has a positive effect on the immunological biomarkers associated with atopic dermatitis. Further our hypothesis is that the difference between the groups (active and placebo) is noticeable during winter time when the disease is typically worse because of the cold weather. The study aim at scientific publication and is double-blinded and placebo-controlled. Time of the intervention is 6-7 months: intervention starts before the Finnish winter time and ends before the summer.

ELIGIBILITY:
Inclusion Criteria:

* A person aged 18-65, legally competent
* Meets Hanifin & Rajka's criteria for atopic dermatitis in the initial interview and eczema has also appeared regularly in adulthood
* The possibility to commit to the research

Exclusion Criteria:

* Cancer or cancer treatments
* Medication that suppresses the immune system (excluding antihistamines)
* Systemic medicine intended for the treatment of atopic dermatitis (orally or as an injection, other than an antihistamine) or the use of clinical phototherapy in the last 6 months.
* Skin infection (such as a eczema that required antibiotic cream or a parasitic infection, e.g.scabies mite) during the last 6 months
* Atopic dermatitis that required hospitalization in the last 2 years
* Psoriasis or other skin disease affecting the study in addition to atopy
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss (TEWL) | 4 or 7 months
  Transepidermal water loss level at designated places

SECONDARY OUTCOMES:
POEM (Patient Oriented Eczema Measure) | Assessment is done every two weeks by the participant
  POEM points during the study
Need of atopy medicines | 4 or 7 months
  Number of medicine free days
EASI (Eczema Area and Severity Index) | 4 or 7 months
  EASI score
Erythema index | 4 or 7 months
  Erythema index at designated places
Skin pH value | 4 or 7 months
  Skin pH value of designated places
Immunological markers in saliva, skin and blood samples | 4 or 7 months
  Immunological markers, like cytokines, in saliva, skin and blood samples and their expression analyzed from RNA.
Adverse events | Assessment is done every two weeks by the participant
  Adverse events during the trial
NRS itch | Assessment is done every two weeks by the participant
  NRS itch score during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Olli Laitinen, PhD, Principal Investigator — Uute Scientific and Tampere University
Locations (1):
- Uute Scientific Oy, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No